CLINICAL TRIAL: NCT01435720
Title: Phase 1/2 Open-Label, Multiple-Dose, Dose-Escalation Study to Evaluate the Safety and Tolerability of SNS01-T Administered by Intravenous Infusion in Patients With Relapsed or Refractory B Cell Malignancies
Brief Title: Safety and Tolerability Study of SNS01-T in Relapsed or Refractory B Cell Malignancies (Multiple Myeloma, B Cell Lymphoma, or Plasma Cell Leukemia (PCL)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Senesco Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNS01-T-001
Record Dates: First submitted 2011-09-14; First posted 2011-09-19 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse; Mantle Cell Lymphoma in Relapse; Diffuse Large B Cell Lymphoma in Relapse; Other B Cell Lymphoma in Relapse; Plasma Cell Leukemia
Keywords: Multiple myeloma; B cell lymphoma; Hematologic disease; Blood protein disorder; Neoplasm, plasma cell; Mantle Cell Lymphoma; Diffuse Large B Cell Lymphoma; Plasma Cell Leukemia; B cell malignancy
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell; Lymphoma, B-Cell; Hematologic Diseases; Blood Protein Disorders; Neoplasms, Plasma Cell; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): 0.0125 mg/kg
  Interventions: Biological: SNS01-T
- Cohort 2 (Experimental): 0.05 mg/kg
  Interventions: Biological: SNS01-T
- Cohort 3 (Experimental): 0.2 mg/kg
  Interventions: Biological: SNS01-T
- Cohort 4 (Experimental): 0.375 mg/kg
  Interventions: Biological: SNS01-T

INTERVENTIONS:
Biological: SNS01-T — 0.05 mg/kg twice weekly x 6 weeks
  Arms: Cohort 2
Biological: SNS01-T — 0.2 mg/kg twice weekly x 6 weeks
  Arms: Cohort 3
Biological: SNS01-T — 0.375 mg/kg twice weekly x 6 weeks
  Arms: Cohort 4
Biological: SNS01-T — 0.0125 mg/kg twice weekly x 6 weeks
  Arms: Cohort 1

SUMMARY:
The purpose of this study is to determine how well SNS01-T is tolerated by relapsed or refractory multiple myeloma, B cell lymphoma or plasma cell leukemia patients when given by intravenous infusion at various doses.

DETAILED DESCRIPTION:
The main purpose is to test the safety and tolerability of SNS01-T. The first group of patients with relapsed or refractory multiple myeloma, plasma cell leukemia or B cell lymphoma will be given a relatively low dose. If tolerated, a second group will receive a higher dose. If tolerated by the second group, a third and then a fourth group will receive higher doses. Treatment-related adverse events (side effects), changes in vital signs, physical examination, and laboratory values will be monitored. Patients will receive twice weekly infusions for 6 weeks and then will be followed monthly for 6 months. A secondary purpose is to explore whether SNS01-T is an effective treatment for multiple myeloma, B cell lymphoma and plasma cell leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. B cell lymphoma patients must have had their diagnosis confirmed histologically. Plasma cell leukemia (PCL) patients must have peripheral clonal plasma cells >20% of peripheral WBC and >2 x 109/L. Multiple myeloma and PCL patients must have been diagnosed by having met all three of the following IMWG criteria:

   * Clonal bone marrow plasma cells >10%
   * Presence of serum and/or urinary M-protein or, if absent, kappa or lambda serum FLC must be > 10 mg/dl accompanied by an abnormal kappa to lambda ratio (<0.26 or >1.65)
   * Evidence of end-organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically, one or more of the following:

     * Hypercalcemia: serum calcium >11.5 mg/100 mL
     * Renal insufficiency: serum creatinine >2mg/dL
     * Anemia: normochromic, normocytic with a hemoglobin value >2 g/100 mL below the lower limit of normal or a hemoglobin value <10 g/100 mL
     * Bone lesions: lytic lesions, severe osteopenia, or pathologic fractures
2. B cell lymphoma patients must have measurable disease defined as at least one lesion that can be accurately measured for response in at least two perpendicular dimensions. Multiple myeloma patients must have measurable disease defined by the following:

   * Serum M-protein ≥0.5g/dL or urine M-protein ≥ 200 mg/24 hours by protein electrophoresis
   * If neither serum nor urine M-protein meet the criteria above, then kappa or lambda serum FLC must be ≥10 mg/dL accompanied by an abnormal kappa to lambda ratio (<0.26 or >1.65) (Serum FLC should only be used for patients without measurable serum or urine M-protein spike.)
   * If neither of the above criteria are met, the presence of plasmacytomata measurable radiographically (CT, PET or MRI) or by direct measurement.
3. Have relapsed or refractory disease after two or more prior treatment lines, each of which may have consisted of either single or multiple regimens. The investigators will ensure that patients have had the benefit of standard treatments before considering the SNS01-T clinical trial.
4. Be at least 2 weeks beyond the last therapy and have recovered from acute toxicities of prior therapies
5. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
6. Have life expectancy of at least 3 months
7. Be ≥18 years of age and willing to provide written informed consent
8. For women and men of childbearing potential, have used effective contraceptive methods for at least 4 weeks prior to dosing and agree to continue using such methods during the study, and for at least 4 weeks after completing the study
9. For women of childbearing potential, have a negative serum pregnancy test within 24 hours before the initiation of SNS01-T therapy
10. Have an absolute neutrophil count >1,000/mm3
11. Have a platelet count >75,000/mm3
12. Have total bilirubin <2.0 mg/dL
13. Have aspartate aminotransferase and alanine aminotransferase <3 times the upper limit of normal
14. Have serum creatinine ≤3 times the upper limit of normal
15. Have hemoglobin ≥8.0 g/dL

Exclusion Criteria:

1. Have presence of nonsecretory myeloma
2. Have an indolent lymphoma such as follicular lymphoma unless the disease is rapidly progressing
3. Requires renal dialysis
4. Have New York Heart Association Class III-IV heart failure classification
5. Have CNS or leptomeningeal disease
6. Have an active infection or serious comorbid medical condition
7. Be receiving other concurrent anticancer agents or therapies
8. Be receiving other concurrent investigational therapies or have received investigational therapies within 4 weeks of screening or 5 half-lives, if known, whichever is shorter
9. Be eligible to receive any other standard therapy available that is known to extend life expectancy
10. Be currently receiving steroids unless equivalent to 20 mg of prednisone or less
11. Be receiving or have received heparin therapeutically within two days before and after treatment with SNS01-T
12. Be pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Week 6
  Safety and Tolerability assessed by frequency, severity, and duration of treatment-related adverse events, changes in vitals signs, physical exams and lab values

SECONDARY OUTCOMES:
Profile of pharmacokinetics | 0.5 hours pre-dose and 0.5, 2, 6 and 24 hours post-dose
  Cmax, area under curve, Tmax. Performed on Weeks 1, 3, 6, 10, 14, 18
Explore tumor response | Weeks 3 and 6, and monthly during a 24-week follow-up period
  IMWG criteria, changes in M-protein, etc. for myeloma and plasma cell leukemia; Lymphoma response criteria, CT/PET scans for B cell lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: John A Lust, MD, PhD, Principal Investigator — Mayo Clinic
Locations (7):
- United States (5):
  - The University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Fred Hutchinson Cancer Research Center/University of Washington Medical Center, Seattle, Washington
  - West Virginia University Mary Babb Randolf Cancer Center, Morgantown, West Virginia
- South Africa (2):
  - Unversity of Cape Town - Groote Schuur Hospital, Cape Town
  - Pretoria East Hospital, Pretoria